CLINICAL TRIAL: NCT03999307
Title: Evaluation of Low-Level Laser Therapy (LLLT) and Flapless Corticopuncture Effect on Accelerating Implant-Supported En-Masse Retraction of the Six Maxillary Anterior Teeth (Clinical Randomized Controlled Trial)
Brief Title: Low-Level Laser Therapy and Flapless Corticopuncture Effect on Accelerating Six Maxillary Anterior Teeth Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-04-2020
Record Dates: First submitted 2019-06-10; First posted 2019-06-26 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: Orthodontic Tooth Movement Acceleration
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Level Laser Therapy (LLLT) (Experimental): In the LLLT group, a low-level laser with wavelength of 808 nm, output of 250 mW, energy of 4 Joules per point and application time of 16 seconds per point will be applied on each tooth of the six maxillary anterior teeth according to this protocol: the root will be divided theoretically into 2 halves; gingival and cervical, and laser will be applied in the center of each half from both buccal and palatal sides which means 4 application points and a total energy of 16 Joules per tooth.
  Interventions: Radiation: Low-Level Laser Therapy (LLLT)
- Flapless Corticopuncture (Experimental): In the flapless corticopuncture group, 3 interdental punctures located between the roots of the six maxillary anterior teeth from both the buccal and palatal sides, will be done using a 1-mm diameter round surgical Tungsten bur with 1 mm depth and 1.5 mm space between each puncture. These punctures start 2 mm from the free gingiva. Besides, an additional 2 parallel set of punctures with the same dimensions of the interdental ones will be done in the extraction sockets from both the buccal and palatal sides.
  Interventions: Procedure: Flapless Corticopunture
- Control (Experimental): Patients in control group will undergo typical orthodontic treatment only with no LLLT or flapless corticopuncture application.
  Interventions: Other: Control

INTERVENTIONS:
Radiation: Low-Level Laser Therapy (LLLT) — LLLT will be applied in this group
  Arms: Low-Level Laser Therapy (LLLT)
Procedure: Flapless Corticopunture — Small holes in the cortical bone will be achieved using 1-mm diameter round surgical Tungsten bur
  Arms: Flapless Corticopuncture
Other: Control — Typical orthodontic treatment with no LLLT or flapless corticopuncture
  Arms: Control

SUMMARY:
The long time needed for orthodontic treatment is considered one of the biggest obstacles that make patients refuse to undergo orthodontic treatment. It also has many disadvantages including higher caries rates, gingivitis, and root resorption. Therefore, the purpose of this study is to evaluate the efficiency of two new noninvasive methods (Low-Level Laser Therapy and Corticopuncture) in accelerating orthodontic tooth movement for the implant supported En-Masse retraction of the six maxillary anterior teeth.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial with a 1:1:1 allocation ratio. Sample size was calculated using Minitab version 15. 36 Participants recruited from patients attending the Department of Orthodontics and Dentofacial Orthopedics at Damascus University with class II division 1 malocclusion that indicates the extraction of first maxillary premolars will be randomly assigned into one of three groups: Low-Level Laser Therapy (LLLT) group, flapless corticopuncture group, or control group. Titanium mini-implants (1.6 mm diameter and 7 mm length) will be inserted between the maxillary second premolar and first molar at approximately 8-10 mm height above the archwires below the mucogingival junction. After complete leveling and alignment of the maxillary dental arch, which will be defined by passive insertion of 19*25 inch S.S. archwire, the retraction stage of the six maxillary anterior teeth will begin.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between (18 - 24) years.
2. Class II Division 1 malocclusion that indicates extraction of two maxillary first premolars with the following parameters:

   ANB: 5 to 10 degrees. Overjet: 5 to 10 mm. Growth Pattern: normal or slightly vertical.
3. All upper teeth are existed (Except for third molars).
4. Mild to moderate crowding (3 mm or less).
5. Patient dose not undergo any medical treatment that interfere with orthodontic tooth movement (Cortisone, NSAIDs, …).
6. Good oral hygiene (Plaque index < 1).

Exclusion Criteria:

1. Any medical condition affecting orthodontic tooth movement.
2. Poor oral hygiene (Plaque index > 1).
3. Patient did not undergo previous orthodontic treatment.
4. Patient lack of commitment toward follow-up appointments.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Duration of en-masse retraction of the six maxillary anterior teeth | The months required to complete the retraction procedure will be recorded, which is expected to be occur within four months
  Assessment will be performed by calculating the time required from the beginning of the six maxillary anterior teeth retraction till the completion of this procedure
Rate of en-masse retraction of the six maxillary anterior teeth | The calculation of the rate of retraction will be done once the retraction procedure has finished which is expected to occur within four months
  Assessment will be performed on study models by dividing the distance that the six maxillary anterior teeth moved during retraction to the time required to retract them to their ideal positions.

SECONDARY OUTCOMES:
Maxillary first molar anchorage loss | This outcome will be measured one day before upper incisors' retraction initiation (T0) and immediately after the completion of retraction (T1) which is expected to occur in 4 months
  Assessment will be performed on study casts by calculating the amount of mesial drifting of the maxillary molar (if any) in millimeters before and after retraction
Root resorption | A CBCT image will be taken one day before the six maxillary incisors retraction initiation (T0) and immediately after the completion of retraction (T1) which is expected to occur in 4 months
  Assessment will be performed by subtracting the root length of each maxillary anterior tooth after retraction from its length before starting retraction procedure.
Changes in the gingival indices | This outcome will be measured one day before the six maxillary incisors retraction initiation (T0) and immediately after the completion of retraction (T1) which is expected to occur in 4 months
  Assessment will be performed clinically using the WHO probe
Change in tooth vitality (the response of the pulp tissue toward external stimuli) | This outcome will be measured one day before the six maxillary anterior teeth retraction initiation (T0) and immediately after the completion of retraction (T1) which is expected to occur in 4 months
  Tooth vitality will be evaluated for each tooth of the six maxillary anterior teeth using Ethyl Chloride applied by a cotton roll on each tooth, which will indicate negative response (no vitality) or positive response (vital pulp)
Changes in the levels of pain and discomfort | These levels will be assessed at: one day, one week, two weeks, and four weeks following the intervention
  Assessment will be performed using questionnaires that include Visual Analog Scale (VAS) for each question, the scale has a minimum scale of 0 (no pain or discomfort) and a maximum scale of 100 (maximum pain or discomfort).
Change in the Oral Health Related Quality of Life associated with anterior teeth retraction. | The OHIP-14 will be assessed immediately after application, after 1, 7, 14, and 28 days of the six maxillary anterior teeth retraction initiation
  Assessment will be performed using the OHIP-14 questionnaire; which is a questionnaire that include 14 questions regarding different aspects of problems that might be associated with retraction (discomfort, stress, chewing difficulties, ...). the patient could choose the answer from a five-point Likert scale (Never, Hardly ever, Occasionally, Fairly often, Very often)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Moaffak A. AlSayed Hasan, DDS, Msc Ortho, PhD Student, Principal Investigator — PhD Student, Department of Orthodontics and Dentofacial Orthopedics - Faculty of Dental Medicine - Damascus University - Damascus - Syrian Arab Republic; Mowaffak Ajaj, DDS, Msc Ortho, PhD, Study Chair — Assistant Professor, Department of Orthodontics and Dentofacial Orthopedics - Faculty of Dental Medicine - Damascus University - Damascus - Syrian Arab Republic; Omar Hamadah, DDS, Msc, PhD, Study Chair — Assistant Professor, Department of Oral Medicine - Faculty of Dental Medicine - Damascus University - Damascus - Syrian Arab Republic
Locations (1):
- Faculty of Dental Medicine, Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AlSayed Hasan MMA, Sultan K, Hamadah O. Low-level laser therapy effectiveness in accelerating orthodontic tooth movement: A randomized controlled clinical trial. Angle Orthod. 2017 Jul;87(4):499-504. doi: 10.2319/062716-503.1. Epub 2016 Nov 21. PMID 27869476
- [Background] Al-Sibaie S, Hajeer MY. Assessment of changes following en-masse retraction with mini-implants anchorage compared to two-step retraction with conventional anchorage in patients with class II division 1 malocclusion: a randomized controlled trial. Eur J Orthod. 2014 Jun;36(3):275-83. doi: 10.1093/ejo/cjt046. Epub 2013 Jun 20. PMID 23787192
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Hoogeveen EJ, Jansma J, Ren Y. Surgically facilitated orthodontic treatment: a systematic review. Am J Orthod Dentofacial Orthop. 2014 Apr;145(4 Suppl):S51-64. doi: 10.1016/j.ajodo.2013.11.019. PMID 24680025
- [Background] Tuncer NI, Arman-Ozcirpici A, Oduncuoglu BF, Gocmen JS, Kantarci A. Efficiency of piezosurgery technique in miniscrew supported en-masse retraction: a single-centre, randomized controlled trial. Eur J Orthod. 2017 Nov 30;39(6):586-594. doi: 10.1093/ejo/cjx015. PMID 28402521
- [Result] Alfawal AM, Hajeer MY, Ajaj MA, Hamadah O, Brad B. Effectiveness of minimally invasive surgical procedures in the acceleration of tooth movement: a systematic review and meta-analysis. Prog Orthod. 2016 Dec;17(1):33. doi: 10.1186/s40510-016-0146-9. Epub 2016 Oct 24. PMID 27696311
- [Result] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579